CLINICAL TRIAL: NCT02497638
Title: A Randomized, Double Blind, Trial of Metformin and Atorvastatin in Delaying Androgen Deprivation Therapy Among Men With Rising PSA Following Radical Prostatectomy or Radiotherapy: The LIGAND (LIpitor and biGuanide to Androgen Delay) Trial
Brief Title: LIpitor and biGuanide to Androgen Delay Trial
Acronym: LIGAND
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug intervention no longer relevant for the proposed population
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-053
Record Dates: First submitted 2015-06-19; First posted 2015-07-14 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: metformin; atorvastatin; prostate-specific antigen; biochemical recurrence
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin; Biguanides; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin and Atorvastatin (Experimental): Atorvastatin 20 mg once daily until progression with one month run-in of 850 mg metformin once daily, followed by 850 mg twice daily of metformin until progression.
  Interventions: Drug: Metformin; Drug: Atorvastatin
- Placebo (Placebo Comparator): One placebo tablet (corresponding to atorvastatin) once daily until progression, with one month of one placebo tablet (corresponding to metformin) once daily, followed by one placebo tablet twice daily until progression.
  Interventions: Drug: Placebo (corresponding to metformin); Drug: Placebo (corresponding to atorvastatin)

INTERVENTIONS:
Drug: Metformin — One month run-in of 850 mg metformin once daily, followed by 850 mg twice daily of metformin until progression.
  Other Names: biguanide
  Arms: Metformin and Atorvastatin
Drug: Atorvastatin — Atorvastatin 20 mg once daily until progression.
  Other Names: lipitor
  Arms: Metformin and Atorvastatin
Drug: Placebo (corresponding to metformin) — One month of one placebo tablet (corresponding to metformin) once daily, followed by one placebo tablet twice daily until progression.
  Arms: Placebo
Drug: Placebo (corresponding to atorvastatin) — One placebo tablet (corresponding to atorvastatin) once daily until progression.
  Arms: Placebo

SUMMARY:
This study is a randomized trial examining the administration of a combination of biguanide metformin and atorvastatin ("Lipitor") to men who are experiencing rising prostate-specific antigen (PSA) levels, despite having undergone radical therapy (surgery and/or radiation).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Histologically confirmed adenocarcinoma of the prostate
* History of radical therapy (i.e., radical prostatectomy, radiotherapy, brachytherapy or prostatectomy with salvage radiotherapy)
* Serum testosterone levels 8.0 nmol/L (230 ng/dL) or greater
* Not currently undergoing treatment for hyperlipidemia or diabetes mellitus
* LDL-cholesterol levels 5 mmol/L or lower
* HgA1c 6.5% or lower
* PSA levels between 2 and 5 ng/mL

Exclusion Criteria:

* Subjects that have been treated for prostate cancer with any of the following:

  i. Cytotoxic chemotherapy; ii. Hormonal therapy within past 3 years; iii. Oral glucocorticoids; iv. Gonadotropin-releasing hormone (GnRH) analogues (e.g., leuprolide, goserelin, degarelix)
* Past treatment with the 5-α reductase inhibitors finasteride and dutasteride within past 5 years
* Past treatment with drugs with antiandrogenic properties (e.g., flutamide, bicalutamide, ketoconazole, progestational agents) within 6 months prior to screening
* Use of metformin or statins within past 2 years
* Planned or concurrent use of metformin, sulfonylureas, thiazolidinediones or insulin for any reason
* Known hypersensitivity or intolerance to metformin or atorvastatin
* Any clinically significant laboratory abnormalities (e.g., severe renal or hepatic impairment) which in the judgment of the investigator would affect the patient's health or the outcome of the trial
* Any condition associated with increased risk of metformin-associated lactic acidosis (e.g., congestive heart failure defined as New York Heart Association (NYHA) class III or IV, history of any type of acidosis, habitual intake of 4 or more alcoholic beverages per day)
* Abnormal liver function test
* Abnormal organ and marrow function

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression (defined as PSA rise to 10 ng/mL or greater, development of clinically overt metastases) or patient/physician desire for androgen deprivation therapy. | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.

SECONDARY OUTCOMES:
Time to androgen deprivation therapy | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
Time to PSA progression | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
Time to disease progression | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
Body mass index | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
  Relationship between body mass index and response to anti-metabolic and anti-cholesterol therapy
Circulating glycated hemoglobin levels | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
  Relationship between circulating glycated hemoglobin levels and response to anti-metabolic and anti-cholesterol therapy
C-peptide levels | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
  Relationship between C-peptide levels and response to anti-metabolic and anti-cholesterol therapy
Adipokine levels | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
  Relationship between adipokine levels and response to anti-metabolic and anti-cholesterol therapy
LDL/HDL cholesterol levels | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
  Relationship between LDL/HDL cholesterol levels and response to anti-metabolic and anti-cholesterol therapy
Triglyceride levels | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
  Relationship between triglyceride levels and response to anti-metabolic and anti-cholesterol therapy
Incidence of adverse events during administration of metformin and atorvastatin to men with prostate cancer. | From date of randomization until the date of progression or patient/physician desire for androgen deprivation therapy, whichever comes first, assessed up to 36 months.
  Assessment of incidence of adverse events from the administration of metformin and atorvastatin to men with prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hamilton, MD, MPH, FRCSC, Principal Investigator — University Health Network, Toronto; Neil Fleshner, MD, MPH, FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada